CLINICAL TRIAL: NCT02093858
Title: The Mechanism of TCF7L2 and SLC30A8 on Antipsychotic-induced Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, PhD, Central South University
Other Study IDs: RRW
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Metabolic Syndrome
Keywords: Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- olanzapine: 15-25mg/day for 24 weeks

SUMMARY:
Almost all of antipsychotics can induce metabolic syndrome,Genetic factors play a key role in the development of metabolic syndrome,TCF7L2 and SLC30A8 are strongestly correlated with metabolic syndrome.Moreover,Antipsychotics have an effect on the expression of TCF7L2 and SLC30A8 genes.It indicates the variations of TCF7L2 and SLC30A8 play an important part in the development of antipsychotics-induced metabolic syndrome.

DETAILED DESCRIPTION:
* In this study, we will determine the effect of olanzapine on the expression of TCF7L2 and SLC30A8.
* The relationship of the polymorphism of TCF7L2 and SLC30A8 with antipsychotic-induced metabolic syndrome in schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of first episode schizophrenia
* Must be able to swallow tablets
* Take only one antipsychotics

Exclusion Criteria:

* liver or renal or cardiovascular diseases
* pregnant or lactating women
* drug and alcohol dependence

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participants met the Diagnostic and Statistical Manual of Mental Disorder-Fourth Edition (DSM-IV) criteria for first episode schizophrenia.All of the patients and their familier are know of the study and sign the informed consent.
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight and blood glucose | 24 weeks

SECONDARY OUTCOMES:
Change of the blood pressure and blood lipid | 24 weeks

OTHER OUTCOMES:
Change of serum insulin | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wu R Rong, PhD, Principal Investigator — Central South University
Locations (1):
- Mental Health Institute, Changsha, Hunan, China